CLINICAL TRIAL: NCT06156618
Title: The Effect of Nitrate Supplement on the Oral Microbiome, Salivary Pellicle Proteins and Vascular Function of Individuals With Dental Erosion
Brief Title: The Effect of Nitrate Supplement on the Oral Microbiome and Saliva in Dental Erosion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Ant Shepherd, Dr Ant Shepherd, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 334090
Record Dates: First submitted 2023-11-09; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Dental Erosion
MeSH Terms: conditions — Tooth Erosion | interventions — Nitrates

STUDY DESIGN:
Intervention Model Description: this study will be a double blind, randomised design, crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active nitrate (Active Comparator): Arm Description: Nitrate Intervention Arm
  Intervention: Beetroot Juice (BJ) with Nitrate Supplements
  Dosage Form: Liquid Dosage: 70 ml Frequency: Twice daily Duration: Seven days Participants assigned to this arm will receive Beetroot Juice (BJ) containing nitrate supplements. The intervention involves the ingestion of 70 ml of BJ twice daily for a duration of seven days. The BJ are designed to be indistinguishable in taste and appearance, ensuring blinding during the study. This arm is a crucial component of the double-blind, randomized crossover trial investigating the effects of nitrate supplements on oral microbiome recovery, blood pressure, and arterial stiffness in both healthy individuals and those with Dental Erosion. Detailed protocol and participant information available in attached documentation.
  Interventions: Dietary Supplement: Nitrate
- Placebo nitrate (Placebo Comparator): Arm Description: Placebo Intervention Arm
  Intervention: Placebo ( Beetroot Juice depleted from nitrate), Identical to the active nitrate in texture, taste, colour and smell.
  Dosage Form: Liquid Dosage: 70 ml Frequency: Twice daily Duration: Seven days Participants in the placebo intervention arm will receive a liquid placebo consisting of flavored water with discolouring dyes. The placebo is administered in the same manner as the active intervention, with participants ingesting 70 ml twice daily for a duration of seven days. This arm serves as a control group in the double-blind, randomized crossover trial, allowing for a comparison with the effects observed in the Beetroot Juice (BJ) with nitrate supplements arm. The order of treatment (BJ or placebo) is randomly assigned and reversed during the second phase of the study to ensure unbiased results. Detailed protocol and participant information available in attached documentation.
  Interventions: Dietary Supplement: Nitrate

INTERVENTIONS:
Dietary Supplement: Nitrate — The proposed study is part of a PhD educational project and will be a double blind, randomised design, crossover trial for the effect of nitrate supplement on healthy control and people with dental erosion (PwDE). This study aims to explore the effect of nitrate supplement on oral microbiome in WMS and SP and its impact on blood pressure and arterial stiffness in healthy controls and PwDE.

SUMMARY:
Dental erosion happens when teeth lose some of their parts because of acid from the things people eat and/or drink or even from their stomach. It can make their teeth hurt and become sensitive. The mouth has a protective shield called salivary pellicle that helps, and there are some special bacteria called Nitrate-reducing bacteria (NRB) that can be good for the mouth and heart. Eating some fruits and vegetables or drinking beetroot can make these bacteria thrive, which might help the heart and blood pressure. This study wants to see how drinking beetroot juice affects these good bacteria in your mouth for people with healthy teeth and those with erosion. This study aims to find out if drinking beetroot juice can change the saliva and bacteria in the mouth for the better, in people with both healthy teeth and those with dental erosion.

The proposed study is part of a PhD educational project and will be a double blind, randomised design, crossover trial for the effect of nitrate supplement on healthy control and people with dental erosion (PwDE). This study aims to explore the effect of nitrate supplement on oral microbiome in WMS and SP and its impact on blood pressure and arterial stiffness in healthy controls and PwDE.

DETAILED DESCRIPTION:
Upon consent being granted, several samples and measurements will be collected from the participant during this research study spanning over 3 visits.

The proposed study is part of a PhD educational project and will be a double blind, randomised design, crossover trial for the effect of nitrate supplements on healthy control and PwDE. This study aims to explore the effect of nitrate supplements on oral microbiome recovery in whole mouth saliva (WMS) and salivary pellicle (SP) and its impact on blood pressure and arterial stiffness in PwDE and healthy controls. The reason this is coming to the HRA is because we do not have an HTA license at the University of Portsmouth.

This study will assess various biomarkers, including salivary proteins and oral microbiome, vascular function, nitrate-reducing activity of oral bacteria, and oxidative stress markers, to understand the impact of chlorhexidine mouthwash on oral and vascular health in PwDE and healthy individuals. The effect of CHX on the structure and composition of the oral microbiome in healthy and PwDE will be analysed. Furthermore, this study will analyse micro and macrovascular endothelial function changes in both groups (healthy and PwDE groups), linking changes to oral microbial communities and cardiovascular function.

Two groups of participants are required for this study [healthy (n=10) and PwDE (n=10) groups] from volunteer participants from the university of Portsmouth (UoP) who have no signs of or reported medical problems (detailed protocol of recruitment attached). Based on power calculation, 12 individuals will be recruited for each group (healthy and PwDE groups) to account for a 16% drop-out rate.

Participants will be approached to volunteer for the study by the chief investigator and PhD researcher through word of mouth, emails via departmental staff lists, University of Portsmouth Dental Academy (UPDA) updates newsletter, UPDA department meetings and presentations about the study during the UPDA's journal club events. A participant information sheet (PIS) and consent form (see attached forms) will be distributed either via email or by handing out hard copies to those wishing to partake in the research. Participants who have returned their completed consent form will be invited to come to UPDA for further assessment of suitability (visit 1).

The participants who has agreed to take part in this research will be invited to attend the University of Portsmouth Dental Academy, Beatty Building (UPDA) for three consecutive visits. They will be invited to attend the UPDA's dental clinics for their first visit for clinical screening and baseline sampling then for their consecutive sampling visits (2 visits) to attend Spinnaker Building, School of Sport, Health & Exercise Science, University of Portsmouth (SbUoP) for further sampling.

Visit 1 (30 minutes-1 hour): This visit will include clinical screening, consent and baseline samples taken and will take place at UPDA dental clinics. The mouths of participants will be screened for suitability to fit in either of the groups (healthy or dental erosion groups) depending on the presence or absence of dental erosion in their teeth. A scoring system called BEWE will be used which is a simple, reproducible and convenient scoring system that can be used for recording clinical findings of dental erosion. If BEWE score is greater than 8 per extant cumulative score and one score 3 in at least one sextant then this means the participant's mouth shows evidence of dental erosion. If a participant is found to be suitable based upon inclusion/exclusion criteria (see attached detailed protocol), they will be invited to attend further appointments.

A medical history, dental history and two further questionnaires (Diet Questionnaire and Reflux Disease Questionnaire) will be completed with participants to ensure that they are suitable for this research study.

After the oral assessment and completing all forms and questionnaires, participants will be assigned to two groups of participants [healthy (n=10) and dental erosion (n=10) groups]. Within each group, the ten participants will be randomly and blindly assigned to further two subgroups by an independent researcher to receive one of the treatments [Beetroot Juice (BJ) (n=5) and placebo (flavoured water with discolouring dyes) (n=5)] as can be seen in the attached protocol. In the same visit, they will then be invited to come to the science laboratory (Beatty Building, UPDA) for several sample collections. As described in the protocol and participant information sheet, these will include measuring participants' blood pressure and brachial artery endothelium-dependent function. Next, venous blood will be collected via venepuncture from the forearm in 4 mL aliquots. After that, saliva and salivary pellicle from teeth and tongue will be collected.

Then each participant from each subgroup will either receive 14 tubes containing 70 ml each of BJ containing nitrate supplements (n=5) or 14 tubes containing the placebo (flavoured water with discolouring dyes) (n=5) depending on the randomisation process. Both versions of the beetroot juice will be identical in taste and appearance. Participants will be blinded to the active nitrate supplement of interest (BJ). Each group will be instructed to intake each product in a reverse order as shown in (figure 1) which will thoroughly be explained by a member of our research team during this visit (visit 1). Specifically, 5 individuals from each group [healthy (n=10) and PwDE (n=10) groups] will be instructed to intake 70 mL each of BJ containing nitrate supplements twice daily for 7 days with the final tube to be taken the morning before their next visit (visit 2) as shown in figure 1. The other 5 individuals will be instructed to intake 70 mL placebo (flavoured water with discolouring dyes) twice daily for 7 days with the final tube to be taken the morning before visit 2. For standardisation, each participant will also be given the same toothpaste to use throughout the duration of the study.

Visit 2 (30-40 minutes per visit) AND Washout and Reverse treatment:

Seven days after visit 1, participants will be invited to return to the (SbUoP) for visit 2, between 9AM-12PM, with the final dose being taken 2 hours prior to their scheduled appointment time. Upon arrival, same samples will be collected and same measurements will also be recorded as that in baseline (blood pressure, brachial artery endothelium-dependent function, venous blood, saliva and salivary pellicles).

After visit 2, each group of participants will be instructed to undertake a four week wash out period before swapping to using the other nitrate supplement (twice a day) for seven more days. The study will end with a final sampling visit on the seventh day of the other nitrate supplement (visit 3) as shown in figure 1.

Visit 3 (30-40 minutes per visit):

Seven days after switching to the alternative nitrate treatment, participants will be asked to take it twice a day and continue this treatment for an additional seven days (visit 3). Then, on the seventh day of this new nitrate treatment (visit 3), participants will be invited for a final sampling visit with final dose taken 2 hours before the oral assessment, as indicated in Figure 1. Upon arrival, same sample and measurements will be repeated as visits 2. Upon completion of final sample collections (visit 3), this will be the end of volunteer participation.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria A) Healthy volunteers Group

Inclusion Criteria:

1. Be aged 18 to 75 years inclusive
2. Have a minimum of 20 natural uncrowned teeth (excluding 3rd molars) present
3. Give written informed consent
4. Be in good general health and oral health (without active caries lesions, gingivitis, periodontitis.
5. No diseases of the soft or hard tissues of the oral cavity
6. No other oral condition affecting the composition of the oral fluids and presented normal salivary flow (stimulated salivary flow >1 mL/min, unstimulated salivary flow > 0.25 mL/min; salivary pH > 6)
7. Show no evidence of dental erosion or/and active dental caries (with BEWE score ≤8 per extant cumulative score per patient and no clinically visible decayed teeth) B) Dental erosion group Inclusion Criteria

1. Same as above of healthy volunteers (1-6). 2. Show evidence of dental erosion (with BEWE score > 8 per extant cumulative score per patient and one score 3 in a sextant. BEWE is a simple, reproducible and convenient scoring system that can be used with the diagnostic criteria for recording clinical findings and examining dental hard tissues other than for caries, guiding the management of erosive tooth wear.

-

Exclusion Criteria:

1. Smokers, using mouthwash or tongue scrapes.
2. Consumption of beetroot juice in normal diet (This will be determined from responses on the diet form).
3. Diagnosed with alcoholism (or drinking more than four times a week, or consuming at least 40 g in males and 20 g in females per day)
4. Presenting conditions associated with vomiting (e.g. anorexia or bulimia), bruxism and Gastro-oesophageal reflux disease (GORD)
5. Occupations associated with increased risk of erosion, such as swimmers and battery, charging and galvanizing workers.
6. Wearing certain types of dental work on specific teeth (e.g., orthodontic appliances, extensive dental bridges, or recent oral surgery
7. Use of antibiotics three (3) months prior to or during this study
8. Use of any over the counter medications other than analgesics or have a known medical condition or currently taking any medication
9. Pregnant or breastfeeding

8. Participation in another clinical study in the month preceding this study 9. Medical condition which requires pre-medication prior to dental visits/procedures.

10. Participants who have eaten/had anything to drink up to two hours before providing a sample (Two hours prior to the trial, participants will be instructed to eat a self-selected light meal and drink 500 ml of water. No other food or fluid will be allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Identification of salivary proteins via SDS-PAGE Electrophoresis: | December 2024
  SDS-PAGE will be used to identify salivary proteins in saliva and pellicle samples and any potential changes in protein bands at a variety of conditions.
Identification of salivary proteins via Proteomics analysis: | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  will identify a number of salivary proteins in saliva and pellicle samples including prolactin inducible protein (PIP) and zinc-alpha-2 glycoprotein (ZAG)
Microbiome diversity using DNA extraction and 16s ribosomal RNA analysis | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  Saliva and pellicle samples will be used to isolate bacterial DNA which will be quantified using a fluorometric method Results from the DNA sequencing will be directly compared between those individuals classified as showing dental erosion and those healthy participants.

SECONDARY OUTCOMES:
Blood pressure measurement: | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  Blood pressure of the brachial artery will be measured following 30 minutes of seated rest in a quiet room using an automated sphygmomanometer. A total of five successive measurements will be taken, with 1-minute rest between readings, with the mean of the final three measurements will be recorded. The mean of the systolic (SBP), diastolic (DBP) and mean arterial pressure (MAP) measurements will be recorded.
Endothelial function test (Iontophoresis) of brachial artery: | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  Iontophoresis will permit the transdermal delivery of Acetylcholine (Ach) and sodium nitroprusside (SNP) to the volar aspect of the right forearm. These chemicals will be introduced through a process called Iontophoresis. Iontophoresis is a unique test where we use a gentle electrical charge to help specific substances get into your skin. This method is beneficial for carefully delivering therapeutic agents through skin or for diagnostic reasons.
Flow-mediated dilation (FMD) of brachial artery: | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  Brachial artery endothelium-dependent function will be measured using the FMD technique as previously described. FMD represents an endothelium-dependent, largely NO-mediated dilatation of conduit arteries in response to an imposed increase in blood flow and shear stress. A high-resolution ultrasound machine will be used to image the brachial artery in the distal third of the upper arm.
Nitrate-reducing activity of oral bacteria | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  To assess the nitrate-reducing activity of oral bacteria for evaluation of nitrate-reducing activity in oral bacteria through a meticulously outlined sequence of future steps.
Nitrate and nitrite in saliva, plasma via Ozone-based chemiluminescence | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  Blood samples:
  Venous blood will be collected and analysed for NO3- and NO2- content
  Saliva samples:
  The WMS will be collected and analysed for NO3- and NO2- content
Oxidative stress markers and redox-related molecules via ELISA: | Baseline (day -7), post each intervention (i.e. Beetroot juice and placebo) on day 1
  ELISA will be used to identify some common Oxidative stress markers and redox-related molecules such as 3-NO-Tyr in saliva and blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth Academy, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan